CLINICAL TRIAL: NCT06506487
Title: Effectiveness of Doll Therapy in People With Dementia: A Mixed Method Research Study
Brief Title: Effectiveness of Doll Therapy in People With Dementia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Zhenti Cui, PhD Candidate, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LL20240509
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doll Therapy plus Routine Nursing Care (Experimental): Participants in this arm will receive doll therapy sessions in addition to routine nursing care. Doll therapy involves the use of lifelike dolls to provide comfort and reduce behavioral and psychological symptoms in people with dementia. The therapy includes activities such as holding, dressing, and interacting with the dolls under the guidance of trained caregivers. Routine nursing care will include standard care practices without additional non-pharmacological interventions.
  Interventions: Behavioral: Doll Therapy
- Routine Nursing Care (No Intervention): Participants in this arm will receive routine nursing care without any additional interventions. Routine nursing care includes standard care practices as provided in the residential care facilities, focusing on the overall well-being and daily needs of the participants.

INTERVENTIONS:
Behavioral: Doll Therapy — Doll therapy involves the use of lifelike dolls to provide comfort and reduce behavioral and psychological symptoms in people with dementia. The therapy includes activities such as holding, dressing, and interacting with the dolls under the guidance of trained caregivers.
  Arms: Doll Therapy plus Routine Nursing Care

SUMMARY:
This study aims to evaluate the effectiveness of doll therapy in reducing the daily dose of medications (DDM), behavioral and psychological symptoms of dementia (BPSD), and improving the activities of daily living (ADL) in people living with dementia (PLwD) in residential care facilities in China. The study employs a cluster randomized controlled trial design, involving 142 participants from six nursing homes, divided into an intervention group receiving doll therapy plus routine nursing care and a control group receiving routine nursing care alone. Additionally, the study will explore the experiences and perceptions of staff and family caregivers through qualitative research methods to provide a comprehensive understanding of the intervention's impact.

DETAILED DESCRIPTION:
Doll therapy, recognized as a non-pharmacological intervention, involves providing lifelike baby dolls to individuals with dementia to elicit positive emotional responses and behaviors. Despite its potential benefits, evidence supporting its efficacy and acceptability remains limited and inconclusive. This mixed-method research study will conduct a cluster randomized controlled trial to systematically evaluate the effectiveness of doll therapy in reducing the daily dose of medications, mitigating behavioral and psychological symptoms, and enhancing daily living activities among Chinese dementia patients in residential care settings. The trial will involve 142 participants from six nursing homes, randomly assigned to either the intervention group (doll therapy plus routine care) or the control group (routine care only). Quantitative outcomes will be measured using standardized scales for medication use, BPSD, and ADL. In parallel, qualitative data will be collected through interviews with staff and family caregivers to gain insights into their experiences and perceptions of doll therapy. The findings are anticipated to inform best practice guidelines for implementing doll therapy in dementia care.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 65 years old.
* Documented diagnosis of dementia.
* Sufficient manual dexterity to hold or caress a doll.
* Sufficient visual acuity to recognize a doll.
* Must have legal family members or next of kin to sign the consent form.

Exclusion Criteria:

* Individuals with mild dementia who do not accept the doll after two attempts.
* Participants who accept the doll but leave it within two weeks.
* Individuals without the capacity to give informed consent and without a legal representative to provide consent on their behalf.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Daily Dose of Medication (DDM) | 12 weeks
  This primary outcome measure will assess the effectiveness of doll therapy in altering the daily dose of medications (DDM) required by participants. The daily dose of medications includes antipsychotics, antidepressants, anxiolytics, and cognitive enhancers, converted to standardized doses (e.g., chlorpromazine equivalents for antipsychotics, diazepam equivalents for anxiolytics, donepezil equivalents for cognitive enhancers, and defined daily dose (DDD) for antidepressants). The change in medication dosage will be measured and compared between the intervention group (doll therapy plus routine care) and the control group (routine care alone).

SECONDARY OUTCOMES:
Change in Behavioral and Psychological Symptoms of Dementia (BPSD) | 12 weeks
  This secondary outcome measure will evaluate the change in behavioral and psychological symptoms of dementia (BPSD) using the Neuropsychiatric Inventory (NPI-12). This inventory includes 12 domains such as delusions, hallucinations, agitation/aggression, depression, anxiety, and others. The scores will be measured and compared between the intervention and control groups. The NPI-12 scores range from 0 to 144, with higher scores indicating more severe symptoms.
Change in Activities of Daily Living (ADL) | 12 weeks
  This secondary outcome measure will assess the change in activities of daily living (ADL) using the Chinese version of the Barthel Index of ADL. This index measures the functional independence of participants in performing daily activities such as feeding, bathing, dressing, toileting, transferring, and walking. The scores will be measured and compared between the intervention and control groups. The Barthel Index scores range from 0 to 100, with higher scores indicating better functional independence.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenti Cui, Principal Investigator — Social and Preventive Medicine, Malaya University
Locations (1):
- Sias University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared after deidentification. Data will be available to researchers who provide a methodologically sound proposal. Data will be available from 3 months to 5 years following article publication. Requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3 months to 5 years following article publication
Access Criteria: Requestors will need to sign a data access agreement.